CLINICAL TRIAL: NCT03111888
Title: Small Feasibility Study for Evaluating the Clinical Effectiveness of 3D Printing for a Patient-specific Silicone Stent Airway Implant
Brief Title: Evaluating the Clinical Effectiveness of 3D Printing for a Patient-specific Silicone Stent Airway Implant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decision
Sponsor: The Cleveland Clinic (Other)
Collaborators: Custom Orthopaedic Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: gildea0217
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patient-Specific Tracheobronchial Stent (Experimental): Observe and document the ability of a patient-specific tracheobronchial stent to improve a patient's quality of life and symptoms associated with airway stenosis.
  Interventions: Device: Silicone Stent Airway Implant

INTERVENTIONS:
Device: Silicone Stent Airway Implant — The Patient-Specific Tracheobronchial Stent is a silicone stent indicated for use in adults that have stenosis of the airway. The subject device takes a CT scan, thresholds out the airway from the other anatomy, and allows the physician to digitally build the stent to his/her desired dimensions. According to the physician's design, a patient-specific stent can be manufactured using rapid prototyping technology. The patient-specific stent is indicated for use with any rigid bronchoscopy/stent application system that fits the design envelope.

SUMMARY:
The goal of the small feasibility trial is to establish a method, material, and patient-specific design that is superior to what is in use today. The first round of patients are well known to the physician investigator and are familiar with the problem that is being resolved. The end goal of the project is to create a new patient-specific design that will last longer, fit better, and cause less trauma to the airway and the patient.

DETAILED DESCRIPTION:
Subjects will be selected from physician investigator's clinical practice where patients have had failure of current stenting procedures to achieve an adequate clinical outcome. A routine CT scan of the chest is required on all individuals going through the procedure for stent placement (rigid bronchoscopy). The physician investigator will use this CT scan to measure and build a patient-specific stent or modify existing stents to fit the specific need.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Patients must be at least 18 years of age
3. Patients must be able to undergo routine non-contrast CT scans of the chest
4. Patient must be stable for general anesthesia and have an airway amenable to rigid bronchoscopy and stent implantation.
5. The patients must have at least an expected 6 month survival.
6. Patient must be able to maintain standard of care follow-up schedule and have access to standard of care medications and nebulizer machines and/or suction and oxygen as required for primary disease management.
7. Patient must be able to personally provide consent and be able to describe Dyspnea and QOL and other patient-reported outcomes (PROs) required by study design
8. Patient must require a stent that is within the design envelope of the patient-specific stents, as defined by COS

Exclusion Criteria:

1. Patients may be excluded if the disease can be managed by simply removing prior stents or performing more conservative therapies.
2. Chronic anticoagulant therapy that could limit the safety of performing rigid therapeutic bronchoscopy in a timely manner. (I.e. Plavix within one year of drug eluding cardiac stent (DES)or 6 weeks following bare metal coronary stent)
3. Unstable cardiac disease
4. Allergy to silicone
5. Stenting to manage vascular compression syndromes.
6. Multi-drug resistant bacterial or fungal chronic infections
7. Emergent/urgent clinically indicated stent.
8. Chronic/permanent mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Observe the outcomes associated with patient-specific airway implants. | Up to 90 days following treatment
  Measure Quality of Life Index through Baseline Dyspnea Index, a validated survey tool
Observe the outcomes associated with patient-specific airway implants. | Up to 90 days following treatment
  Measure Quality of Life Index through Transitional Dyspnea Index, a validated survey tool

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Gildea, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No